CLINICAL TRIAL: NCT05623111
Title: Perineural Injections of Incobotulinumtoxin-A for Diabetic Neuropathic Pain of the Lower Extremities: A Double-blind, Randomized, Placebo-controlled Study
Brief Title: Perineural Injections of Incobotulinumtoxin-A for Diabetic Neuropathic Pain of the Lower Extremities
Acronym: PINBOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Merz Pharmaceuticals GmbH (Industry); Toyota Foundation Denmark (Unknown); Steno Diabetes Center Zealand Region (Unknown); Shipwright Per Henriksen, R., and wife Foundation (Unknown); The GCP unit at Copenhagen University Hospital (Unknown); Capital Region Pharmacy, Denmark (Unknown)
Responsible Party: Principal Investigator, Bo Biering-Soerensen, Senior Physician, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PINBOT
Record Dates: First submitted 2022-10-31; First posted 2022-11-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 2-armed active/placebo 1:1 ratio
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Incobotulinumtoxin-A (Active Comparator): 100 units of incobotulinumtoxin-A in 5ml of sterile saline around both distal ischial nerves.
  Interventions: Drug: Incobotulinumtoxin-A 100 UNIT Injection
- Placebo (Placebo Comparator): 5ml sterile saline with small amounts of human albumin and sucrose (identical to binding agents in active vials)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Incobotulinumtoxin-A 100 UNIT Injection — Perineural injection
  Arms: Incobotulinumtoxin-A
Drug: Saline — Placebo containing trace amounts of human albumin and sucrose, diluted with 5ml of sterile saline.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test perineural injections (injections around a nerve) of incobotulinumtoxin-A in participants with diabetic nerve pain of the feet and lower legs.

The main questions it aims to answer are:

* Is the treatment safe and effective?
* Does the treatment affect participants quality of life, depression, physical activity, daily life, and sensation?

Participants will be treated every 12 weeks, for a total of 24 weeks, with either incobotulinumtoxin-A or a placebo.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled trial, investigating the safety, efficacy, use of rescue medication, and impact on NPSI scores, health-related QoL, activities of daily living (ADLs) and levels of physical activity of perineural incobotulinumtoxin-A (iBonT-A) or placebo injections, in persons with DNP of the lower extremities.

Participants will be randomly assigned via simple block randomization to receive either 100 units of iBonT-A in each leg (total of 200 units), or a placebo in each leg, injected perineurally around both distal sciatic nerves once every 12 weeks, for a total of 24 weeks.

Injections are performed with sonographic guidance by an experienced operator. Contents of the blinded vials, containing either 100 U of iBonT-A or a placebo consisting of small amounts of sucrose and albumin are diluted in 5 ml of sterile saline. The injection point is just distal to the sciatic nerve bifurcation. The skin is penetrated from the lateral side using a non-cutting needle (Pajunk, SonoBlock, 22G x 80 mm, Facet S Tip). With the needle in plane in relation to the ultrasound probe, the nerves are visualized in short axis. The needle tip is placed inside the common sheath surrounding the tibial and peroneus communis nerves. The location of the needle tip is verified with small boli of sterile saline solution in combination with ultrasound. Correct distribution of the injectant is confirmed with dynamic scanning. Fluid distention must be seen around both components. When confirmation of optimal needle placement the 100 units iBonT-A or placebo is injected. The procedure is repeated for both legs.

Participants will be asked to rate their neuropathic pain once a day, as well as register their daily use of rescue medication. Secondary outcome measures will be rated at baseline and at 4, 12, 16 and 24 weeks.

Safety information consists of adverse events recording, as well as motorfunction and sensory changes over time.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older
* Are diagnosed with diabetes type I or II
* Score 3 or above on the Doleur Neuropathique 4 interview section
* Suffer from pain of the lower extremities which

  * is considered by the participant as their dominant overall dominant pain
  * is rated at least 4 out of 10 of the NRS pain scale in both legs (on average over the past 7 days)
  * is present in both feet, roughly symmetrically.
  * has been present for at least 6 months
* Show sensory deficits and/or allodynia or hyperalgesia in the painful area, consistent with the IASP definition of probable chronic neuropathic pain40.
* Are in a stable analgesic treatment regime for at least 1 month prior to inclusion and for the duration of the study
* Are using an approved, safe contraceptive (for premenopausal women)
* Speak, read, and understand Danish

Exclusion Criteria:

* • Have a known allergy or hypersensitivity to BonT-A

  * Have been treated with BonT in the last 6 months.
  * Are diagnosed with myasthenia, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
  * Have a known malignant condition
  * Have an ongoing infection in the area of injection
  * Are expecting to change their pain medication during the study period
  * Have been treated with topical agents such as capsaicin or lidocaine products in the affected areas for at least 3 months prior to inclusion
  * Are diagnosed with a competing cause of central or peripheral neuropathic pain, or other painful chronic conditions of the lower extremities, such as:

    * spinal stenosis
    * claudication
    * previous trauma or nerve injury
    * cancer related pain
  * Have a psychiatric condition that affects their completion of the study, as assessed by the investigator.
  * Are active abusers of alcohol or illegal substances
  * Are using or receiving treatment with cannabis products of any kind
  * Are pregnant or planning pregnancy during the study period
  * Score more than 12 on the Charlson Comorbidity Index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in daily neuropathic pain scores | Recorded once daily for 1 week prior to first injection and daily for the duration of the study. Outcome is defined as differences in change from baseline of average daily and weekly pain scores between groups.
  Differences in pain scores, as measured by the Numeric Rating Scale (0-11), between groups.

SECONDARY OUTCOMES:
Use of rescue medication | Recorded once daily for 1 week prior to first injection and daily for the duration of the study. Defined as differences in change from baseline of average days per week of rescue medication usage across the study period.
  Recorded using pain diary with simple Yes/No for use of any rescue medication. Changes in use of rescue medication over time and between groups.
Neuropathic Pain Symptom Inventory | Baseline, 4 weeks, 12 weeks, 16 weeks, 24 weeks.
  Changes in NPSI total and sub-scores over time and between groups.
Health-related quality of life | Baseline, 4 weeks, 12 weeks, 16 weeks, 24 weeks.
  EQ-5D-5L
Activities of daily living | Baseline, 4 weeks, 12 weeks, 16 weeks, 24 weeks.
  Canadian Occupational Outcome Measure (COPM)
Physical activity | Baseline, 4 weeks, 12 weeks, 16 weeks, 24 weeks.
  Grimby-Saltin Physical Activity Scale, Danish Version (PAS-2-DK)
Depression symptoms | Baseline, 4 weeks, 12 weeks, 16 weeks, 24 weeks.
  Beck Depression Inventory II (BDI-II)
Adverse events | Number and nature of adverse events compared between groups at 24 weeks.
  Incidence, severity and character of adverse, compared between active and placebo groups
Motorfunction of the lower legs. | Baseline, 4 weeks, 12 weeks, 16 weeks, 24 weeks.
  Oxford MRC Muscle Power Assessment
Sensory function | Baseline, 4 weeks, 12 weeks, 16 weeks, 24 weeks.
  Sensation of the lower legs and feet, as measured by Quantitative Sensory Testing, according to the DFNS protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Biering-Sørensen, MD, Study Director — Neurological Pain Clinic, Rigshospitalet
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Study data will be published in anonymised format as supplementary material to publications. Study protocol, SAP, ICH And analytic code available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be published as supplementary material to publications.
Access Criteria: Open Access

REFERENCES:
- [Derived] Klee M, Hormann Thomsen T, Enggaard TP, Bitsch MS, Simonsen L, Jensen RH, Biering-Sorensen B. Perineural injections of incobotulinumtoxin-A for diabetic neuropathic pain of the lower extremities: protocol for a phase II, single-centre, double-blind, randomised, placebo-controlled trial (the PINBOT study). BMJ Open. 2024 Jan 22;14(1):e074372. doi: 10.1136/bmjopen-2023-074372. PMID 38262642